CLINICAL TRIAL: NCT06113029
Title: Prevalence of Depressive Disorders and Anxiety Disorders Among Sample of Patients With Chronic Liver Disease Attending Assiut University Hospitals.
Brief Title: Depressive and Anxiety Disorders in Patients With Chronic Liver Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Ashraf Mohamed Badr, Principal investigator, Assiut University
Other Study IDs: Depression and liver
Record Dates: First submitted 2023-10-26; First posted 2023-11-02 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; liver
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Participants not known to have neither chronic liver diseases nor Psychiatric disorders
  Interventions: Diagnostic Test: The Hamilton Rating Scale for Anxiety; Diagnostic Test: The Beck Depression inventory; Diagnostic Test: Rand SF-36 Questionnaire
- Diseased group: Participants known to have chronic liver diseases
  Interventions: Diagnostic Test: The Hamilton Rating Scale for Anxiety; Diagnostic Test: The Beck Depression inventory; Diagnostic Test: Rand SF-36 Questionnaire

INTERVENTIONS:
Diagnostic Test: The Hamilton Rating Scale for Anxiety — The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Diagnostic Test: The Beck Depression inventory — one of the most widely used instruments for measuring the severity of depression
Diagnostic Test: Rand SF-36 Questionnaire — The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). All scales do contribute in different proportions to the scoring of both PCS and MCS measures

SUMMARY:
The aim of this observational study is to learn about the prevalence of depressive and anxiety disorders among patients with chronic liver diseases

DETAILED DESCRIPTION:
Major depressive disorder (MDD), or clinical depression, is a psychiatric disorder characterized by 2 or more weeks of persistently depressed mood accompanied by symptoms such as feelings of worthlessness, guilt, hopelessness, helplessness, loss of self-esteem, sleep disturbance, changes in oral intake, anhedonia, loss of interest, and suicidality. The american psychiatric association, on the definition of anxiety, describes anxiety as the anticipated anticipation of a future danger or negative event, accompanied by feelings of dysphoria or physical symptoms of tension. The elements exposed to risk may belong both to the internal world and to the external world. depression is highly prevalent globally and is a leading cause of disability. The global burden of disease study found depression to be a leading cause of disability among all illnesses. Liver cirrhosis is one of the diseases commonly associated with depression.chronic liver disease is the progressive destruction and regeneration of the liver parenchyma leading to fibrosis and cirrhosis (normally lasts 6 months). The etiologic agents of CLD include hepatotropic viruses (HBV and HCV), fatty liver, alcohol, autoimmune hepatitis, etc. The mortality of CLD patients remains high not only due to irreversible cirrhosis, but also multiple complications such as HCC and mental disease, especially depression. The progressive nature of this disease results in high rates of hospitalization, extensive exposure to medications, increased financial burden, frequent need for invasive procedures, changes in body image, and an increase in morbidity and mortality. All these factors contribute to the physical and psychological stress that mediates the development of depressive symptom high rates of depression have been documented in patients with decompensated liver disease and in those anticipating liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. patients admitted or attending at Rajhi university hospital with chronic liver disease including: viral (hepatitis B and C), autoimmune (primary biliary cirrhosis, primary sclerosing cholangitis and autoimmune hepatitis), non-alcoholic steatohepatitis, Morbus Wilson and cryptogenic CLD.
2. age group above 18 years old.

Exclusion Criteria:

1. patients with chronic liver disease with other psychiatric disorders other than depression and anxiety.
2. patients with acute complication of chronic liver disease.
3. patients with chronic liver disease who underwent liver transplation.
4. patients with chronic liver disease under antiviral therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver diseases
Sampling Method: Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experienced depressive or anxiety disorders | Baseline
  Each participant will be asked to fill items of questionnaires like The Beck Depression inventor, The Hamilton Rating Scale for Anexity and Rand SF-36 Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Salma Ashraf Mohamed Badr, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Vahia VN. Diagnostic and statistical manual of mental disorders 5: A quick glance. Indian J Psychiatry. 2013 Jul;55(3):220-3. doi: 10.4103/0019-5545.117131. No abstract available. PMID 24082241
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Huang X, Liu X, Yu Y. Depression and Chronic Liver Diseases: Are There Shared Underlying Mechanisms? Front Mol Neurosci. 2017 May 8;10:134. doi: 10.3389/fnmol.2017.00134. eCollection 2017. PMID 28533742